CLINICAL TRIAL: NCT06891339
Title: The Effect of a Patient-oriented Mobile Application Used by Laparoscopic Cholecystectomy Patients in the Perioperative Period on Anxiety, Complications, Comfort and Satisfaction.
Brief Title: The Effect of Mobile Application Used by Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, İmren Erer, Msc, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Laparoscopic cholecystectomy; imren erer (Registry Identifier: The effect of a mobile application used by patients)
Record Dates: First submitted 2025-03-13; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Surgical Patient; Nursing Caries; Laparoscopic Cholecystectomy
Keywords: Laparoscopic cholecystectomy, surgical patient, nursing care
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Experimental Group:
  Patients will receive information about the mobile app and install it for free. Preoperative education, pain monitoring, and complication tracking will be conducted via the app. Video consultations will be available for wound care.
  On surgery day, they will receive standard care. Anxiety will be assessed on postoperative day 1, and daily follow-ups will continue until day 7, when they will complete the Comfort Scale, Patient Satisfaction Questionnaire, and State Anxiety Inventory via the app.
  Control Group:
  Patients will receive standard care. Anxiety will be assessed on day 1. They will be informed about a day 7 follow-up call and provided with VAS pain scales and complication checklists.
  On day 7, a phone interview will collect responses to the Comfort Scale, Patient Satisfaction Questionnaire, and State Anxiety Inventory, along with hospital readmission details.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effect of a patient-oriented mobile application (Experimental): Experimental Group:
  Patients will receive information about the mobile app and install it for free. Preoperative education, pain monitoring, and complication tracking will be conducted via the app.
  Video consultations will be available for wound care. On surgery day, they will receive standard care. Anxiety will be assessed on postoperative day 1, and daily follow-ups will continue until day 7, when they will complete the Comfort Scale, Patient Satisfaction Questionnaire, and State Anxiety Inventory via the app.
  Interventions: Other: mobile application
- standard care (Experimental): Control Group:
  Patients will receive standard care. Anxiety will be assessed on day 1. They will be informed about a day 7 follow-up call and provided with VAS pain scales and complication checklists.
  On day 7, a phone interview will collect responses to the Comfort Scale, Patient Satisfaction Questionnaire, and State Anxiety Inventory, along with hospital readmission details.
  Interventions: Other: mobile application

INTERVENTIONS:
Other: mobile application — The aim is to evaluate whether a patient-centered mobile application with smartphone-based systematic follow-up assessment during the perioperative period can improve surgery-related anxiety, complications, comfort, and patient satisfaction compared to standard care. This thesis will be one of the pioneering studies in this field.
  Other Names: standard care

SUMMARY:
The aim of this study is to evaluate whether a patient-centered mobile application used during the perioperative period can improve anxiety, complications, comfort, and patient satisfaction compared to standard care.

DETAILED DESCRIPTION:
Surgical intervention is a life-threatening condition. It is known that fear and anxiety experienced throughout the surgical process disrupt homeostatic balance, leading to biological, psychological, and social problems in individuals and prolonging the length of hospital stay.

In surgical cases that typically require a hospital stay of one day or less, when there is insufficient time for proper education and guidance, patients may experience anxiety and difficulties. This can lead to repeated hospital visits and increased costs. Effective and accurate communication between the patient and the nurse can ensure the best implementation of nursing care, help the patient feel safer, reduce anxiety, increase care satisfaction, and lower costs.

Complications frequently arise after hospital discharge. Due to a lack of information regarding recovery expectations, many patients may feel insecure, anxious, and alone.

The use of the internet for health information has significantly increased over the past decade. Mobile medical applications can be a useful tool for improving perioperative patient education and care. Most acute care hospitals provide discharge instructions in the form of a brochure, which is often difficult to follow. A mobile application could serve as an educational and instructional resource for patients throughout the perioperative period. It can provide real-time feedback on patients' adherence to perioperative ERAS elements and demonstrate their ability to aid recovery.

There are very few studies investigating the ability of mobile applications to assist in the recovery of surgical patients. Various studies have shown that complications, pain, anxiety, unexpected primary care visits, hospital readmissions, and rehospitalizations are primarily caused by a lack of information.

The aim of this study is to evaluate whether a patient-centered mobile application used during the perioperative period can improve anxiety, complications, comfort, and patient satisfaction compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

Having a smartphone to install the mobile application No barriers to communication in Turkish Scheduled for surgery Willing to participate in the study Above 18 years of age Sufficient ability to use the mobile application

Exclusion Criteria:

Communication barriers Inability to use the mobile application Unwillingness to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-09-16 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The effect of a patient-oriented mobile application used by laparoscopic cholecystectomy patients in the perioperative period on anxiety, complications, comfort and satisfaction. | 2 months
  To evaluate whether it can improve patients' concerns, complications, comfort, and patient satisfaction regarding surgery.

IPD SHARING:
Plan to Share IPD: No
The data of the study will be stored for 5 years.

REFERENCES:
- [Background] Bertocchi E, B. G. (2023, October 11). iColon, a Patient-focused Mobile Application for Perioperative Care in Colorectal Surgery: Results from 444 Patients. Journal of Telemedicine and Telecare, 11(1). Bertocchi, E., Barugola , G., Gentile, I., Zuppini, T., & Zamperini, M. (2021, November). iColon, a patient-focused mobile application for perioperative care in colorectal surgery: an observational, real-world study protocol. BMJ open, 11(11). Carlier, J. R.-G. (2021). Pain Evaluation after Day-Surgery Using a Mobile Phone Application. Anaesthesia, Critical Care & Pain Medicine, 40(3). Dönmez, E., Dolu, İ., & Yılmaz, Ş. (2022). VALIDITY AND RELIABILITY OF A QUESTIONNAIRE TO MEASURE THE PATIENT SATISFACTION WITH NURSING CARE QUALITY TURKISH VERSION. Asia Pacific Journal of Health Management, 17(2). Jaensson, M. D. (2017). Evaluation of Postoperative Recovery in Day Surgery Patients Using a Mobile Phone Application: a Multicentre Randomized Trial. British Journal of Anaesthesia, 119(5), s. 1030-1038. Ko, Y. H. (2021, March 21). The Development of a Mobile Application for Older Adults for Rehabilitation Instructions After Hip Fracture Surgery. Geriatric Orthopaedic Surgery & Rehabilitation, 12(2). Li, C. H. (2019). Monitoring of Home Recovery Using the 317-Nursing Mobile Application Following day-case Surgery in Children: Perspectives from both Nurses and Patients. NIH, 98(31). Morte, K., Marenco , C., Lammers, D., Bingham, J., Sohn, V., & Eckert, M. (2021). Utilization of Mobile Application Improves Perioperative Education and Patient Satisfaction in General Surgery Patients. American Journal of Surgery, 221(4), s. 788-792. Noel, W., Bosc, R., Jabbour, S., Keçiçyan, E., Hersant, B., & Meningaud, J.-P. M. (2017). Smartphone-Based Patient Education in Plastic Surgery. Annals of Plastic Surgery, 79(6), s. 529-531. Özyürek, H., & Göktaş, S. (2021). Acil ve Elektif Cerrahide Hastaların Anksiyete Düzeylerinin ve Hemşirelik Bakım Memnuniyetlerinin Değerlendirilmesi. Sağlık Bilimleri Üniversitesi Hemşirelik Dersgisi, 3(2), s. 83-92. Ponder, M. V.-Y. (2021). Mobile Health Application for Patients Undergoing Breast Cancer Surgery: Feasibility Study. JCO Oncology Practice, 17(9). Yeşilot, S. B., Çiftçi, H., & Yener, M. K. (2021). Lokal Anestezi Altında Lipom Eksizyonu Yapılan Bireylerde Stres Küpü ile Dikkati Başka Yöne Çekme Uygulamasının Ağrı ve Anksiyete Üzerine Etkisi: Randomize Kontrollü Deneysel Çalışma. Ege Tıp Dergisi, 60(3), 219-229. Özsoy, F., Yıldız, M., Gülücü, S., & Kulu, M. (2018). Doğum ağrısı ve bazı psikiyatrik özel-likler arasındaki ilişki. KSU Medical Journal, 13(2), 43-47.